CLINICAL TRIAL: NCT03365869
Title: A Phase Ⅱ Pilot-Study With Sirolimus for the Treatment of Systemic Sclerosis
Brief Title: A Pilot-Study of Sirolimus for the Treatment of Systemic Sclerosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PKUPH-R-SRL
Record Dates: First submitted 2017-12-04; First posted 2017-12-07 (Actual); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Systemic | interventions — Sirolimus

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sirolimus (Active Comparator): Add sirolimus according to the protocol. Sirolimus active: 2mg po. QD
  Interventions: Drug: Sirolimus
- placebo (Placebo Comparator): sirolimus placebo: 2mg po. QD
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus — Sirolimus or placebo were added to patients every day
  Other Names: placebo

SUMMARY:
The purpose of the study is to examine the safety and effectiveness of sirolimus treatment for people with systemic sclerosis.

The investigators perform a multi-centre, double-blind pilot trial with sirolimus in SSc.The investigators evaluate the effectiveness and safeness of sirolimus for Systemic Sclerosis by randomized controlled study (sirolimus 2mg/d (N = 36) versus placebo group (N = 36)).

DETAILED DESCRIPTION:
Each SSc patients (n=72) received sirolimus or placebo (active group: placebo group =1:1, 2mg/day， oral administration, (SIR 2mg, po., Qd) .

The end points were the changement of modified RSS and the adverse events or severe adverse events onset.

ELIGIBILITY:
Inclusion Criteria:

* Meet the American College of Rheumatology criteria for the diagnosis of SSc, 2013.
* Disease duration less than 5 years.
* mRSS was under stable level (>1 month) at the time inclusion.
* Negative urine pregnancy test
* Written informed consent form

Exclusion Criteria:

* Diagnosed with localized scleroderma .
* Added with immunosuppressor in one month such as MTX, AZA, CYC.
* Added with anti-fibosis drug in one month.
* Prednisone >10mg QD before inclusion.
* Sever chronic liver, kidney, lung or heart dysfunction; (heart failure (≥ grade III NYHA), hepatic insufficiency (transaminases> 3N) )
* Serious infection such as bacteremia, sepsis
* Mental disorder or any other chronic illness or drug-abuse that could interfere with the ability to comply with the protocol or to give information
* Cancer or history of cancer cured for less than five years (except in situ carcinoma of the cervix or Basocellular carcinoma)
* Positive HIV test
* Positive urine pregnancy test
* Combined with the other connective tissue diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2018-06-01 (Estimated); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants whose modified Rodnan skin score （mRSS）decreasing | week 48
  mRSS was evaluated in 17 sites of skin.

SECONDARY OUTCOMES:
The number of adverse event and severe adverse event occured | week 48
  SAE were recorded as life-threatening and others were AE.

CONTACTS AND LOCATIONS:
Overall Officials: Mu Rong, Poster, Principal Investigator — Peking University Institute of Rheumatology and Immunology